CLINICAL TRIAL: NCT00794469
Title: Water Induced Thermogenesis in Obese Children
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Eden Springs (Unknown)
Responsible Party: Gal Dubnov-Raz, Hadassah Medical Organization
Other Study IDs: GDR-HMO-CTIL
Record Dates: First submitted 2008-11-19; First posted 2008-11-20 (Estimated); Results first posted 2009-11-25 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2008-11

CONDITIONS: Obesity
Keywords: Resting metabolic rate
MeSH Terms: conditions — Obesity | interventions — Water

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Water: obese children (body mass index > 95th percentile for age and sex) that will drink cold water
  Interventions: Other: Water

INTERVENTIONS:
Other: Water — Children will drink 10 cc/kg of cold water(4 degrees centigrade)

SUMMARY:
Drinking water is largely advocated for obesity prevention and management. Recent studies have suggested that water has a thermogenic effect, this has not been examined in children. In this study, we will measure the resting metabolic rate of 21 obese children before, and during drinking cold (4 degrees centigrade)water for up to 60 minutes.

ELIGIBILITY:
Inclusion Criteria:

* obesity
* agreement and informed consent

Exclusion Criteria:

* non-agreement

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: obese children participating in a lifestyle education and weight management program.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2008-12; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Optimal Sport Medicine Center, Jerusalem, Israel

REFERENCES:
- [Background] Boschmann M, Steiniger J, Hille U, Tank J, Adams F, Sharma AM, Klaus S, Luft FC, Jordan J. Water-induced thermogenesis. J Clin Endocrinol Metab. 2003 Dec;88(12):6015-9. doi: 10.1210/jc.2003-030780. PMID 14671205

RESULTS

PARTICIPANT FLOW:
Groups:
- Water: obese children (body mass index >95th percentile for age and sex) that will drink 10cc/kg of cold water (4 degrees centigrade)
Period: Overall Study
Arm/Group | Water
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Water
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 9.8 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 11
Region of Enrollment [Number; unit: participants]
  Israel | 21
resting metabolic rate [Mean (Standard Deviation); unit: kcal/d] — resting metabolic rate
  kcal/d | 1109 (385)

OUTCOME MEASURES:

1. Primary Outcome: Post-drinking Metabolic Rate
Description: resting metabolic rate after drinking water
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: kcal/d
Arm/Group | Water
Number analyzed (Participants) | 21
kcal/d | 1487 (277)

2. Primary Outcome: Baseline Metabolic Rate
Description: baseline metabolic rate
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: kcal/d
Arm/Group | Water
Number analyzed (Participants) | 21
kcal/d | 1109 (385)

ADVERSE EVENTS:
Arm/Group | Water
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No